CLINICAL TRIAL: NCT04069962
Title: The Effectiveness of Patient Coaching Within the Comprehensive Geriatric Assessment Process on Quality of Life in Older Patients With Cancer Receiving Systemic Therapy: a Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of CGA on QoL in Older Patients With Cancer Receiving Systemic Therapy
Acronym: G-oncoCOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: s62123
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Geriatrics; Comprehensive Geriatric Assessment
Keywords: cancer; older persons; comprehensive geriatric assessment; geriatric interventions; patient compliance
MeSH Terms: conditions — Neoplasms; Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the control group will receive CGA coordinated by the oncology team as standard of care, including geriatric recommendations for interventions communicated to the treating physician (eg. referral to the social worker, psychologist, dietician).
- Intervention group (Experimental): Patients in the intervention group, the CGA including geriatric recommendations for interventions will be coordinated by the geriatric team and will be complemented with patient coaching.
  Interventions: Behavioral: CGA coordination by geriatric team including intensive patient coaching and follow-up

INTERVENTIONS:
Behavioral: CGA coordination by geriatric team including intensive patient coaching and follow-up — In the intervention group, the CGA including geriatric recommendations for interventions will be coordinated by the geriatric team and will be complemented with patient coaching. This intervention aims to support patient empowerment by improving self-efficacy and supporting self-management of existing age-related problems before systemic therapy or occurring during systemic therapy, and includes an individual counselling session at start of systemic therapy to discuss the recommendations with the patient and to determine their priorities.
  Arms: Intervention group

SUMMARY:
The G-oncoCOACH study aims to evaluate the effectiveness of the Comprehensive Geriatric Assessment (CGA) process coordinated by a geriatric team in combination with intensive patient coaching compared to the current standard of care, which is CGA coordinated by an oncology team.

DETAILED DESCRIPTION:
The G-oncoCOACH study aims to evaluate the effectiveness of the Comprehensive Geriatric Assessment (CGA) process coordinated by a geriatric team in combination with intensive patient coaching compared to the current standard of care, which is CGA coordinated by an oncology team. The Medical Research Council (MRC) Framework, developed to test complex interventions, is used to design this study. A multicenter randomized controlled trial will be conducted in two academic hospitals (UZ Brussel - UZ Leuven) with a follow-up at 3, 6 and 12 months after the start of systemic therapy. Patients will be recruited in both academic hospitals in the period between the cancer diagnosis and the start of the systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 70 years and older
* diagnosis of cancer (solid tumors)
* starting systemic therapy (chemotherapy, immunotherapy, targeted therapy or hormonal therapy)

  * curative intent (neo-adjuvant / adjuvant / concomitant / other)
  * palliative intent (first line / second line)
* patients must be able to comply with the study procedures
* physician-estimated life expectancy must be more than 6 months

Exclusion Criteria:

* patients with antihormonal monotherapy
* previous participation in geriatric intervention studies
* patients included in clinical trials with non-registered anticancer drugs

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL): EORTC QLQ-C30 | QoL at 6 months since the start of the systemic therapy
  QoL measured by the EORTC Qlq - C30. HRQOL evaluation was performed using the European Organization for Research and Treatment Quality of Life Questionnaire core 30 (EORTC QLQ-C30) Global Health Status Scale (GHS). The two general questions 29 and 30 are selected: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?". Patients answer these two questions by means of seven-point Likert scales and the two scores are combined to define the GHS. The GHS score is linearly transformed to a 0-100 score to facilitate statistical interpretation. A higher HRQOL is reported by a higher GHS score.

SECONDARY OUTCOMES:
QoL: EORTC QLQ-C30 | QoL at 3 and 12 months since the start of the systemic therapy
  QoL measured by the EORTC Qlq - C30. HRQOL evaluation was performed using the European Organization for Research and Treatment Quality of Life Questionnaire core 30 (EORTC QLQ-C30) Global Health Status Scale (GHS). The two general questions 29 and 30 are selected: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?". Patients answer these two questions by means of seven-point Likert scales and the two scores are combined to define the GHS. The GHS score is linearly transformed to a 0-100 score to facilitate statistical interpretation. A higher HRQOL is reported by a higher GHS score.
Evolution in QoL: EORTC QLQ-C30 | over 1 year follow up since the start of the systemic therapy
  QoL measured by the EORTC Qlq - C30. HRQOL evaluation was performed using the European Organization for Research and Treatment Quality of Life Questionnaire core 30 (EORTC QLQ-C30) Global Health Status Scale (GHS). The two general questions 29 and 30 are selected: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?". Patients answer these two questions by means of seven-point Likert scales and the two scores are combined to define the GHS. The GHS score is linearly transformed to a 0-100 score to facilitate statistical interpretation. A higher HRQOL is reported by a higher GHS score.
Measurement of patient satisfaction: questionnaire | over 1 year follow up since the start of the systemic therapy
  Self-constructed questionnaire on patient satisfaction measuring the satisfaction of the patient with the care that has been received since the start of the systemic treatment (using a 5-point Likert scale; range 1 (not satisfied at all) -5 (very satisfied))
Evolution of functional status (FS) measured by Activities of Daily Living (ADL) | over 1 year follow up since the start of the systemic therapy
  FS measured by Activities of Daily Living (ADL). The ADL scale includes six items (bathing, dressing, toileting, transferring, continence and feeding), with a score for each item scores ranging from one (able to perform the activity) to four (unable to perform the activity) (range: 6-24).
Evolution of functional status (FS) measured by Instrumental Activities of Daily Living (IADL) | over 1 year follow up since the start of the systemic therapy
  FS measured by Instrumental Activities of Daily Living (IADL). The Lawton scale includes eight items (ability to use the telephone, shopping, cooking, housekeeping, doing laundry, taking own medication, making transports and ability to handle finances), with a score for each item of zero (low function, dependent) or one (high function, independent). Because some of these items (cooking, housekeeping and doing laundry) are only fully applicable in women, these three items were not assessed in males in the original form, so the total score in men ranged from zero to five (range women: 0-8; range men: 0-5).
Rate of falls | at 3, 6 and 12 months since the start of systemic therapy
  Rate of falls measured by self-report of fall history
Measurement of systemic therapy-related adverse events | over 1 year follow up since the start of the systemic therapy
  Measurement of systemic therapy-related adverse events based on the NCI Common Terminology Criteria for Adverse Events, NCI CTCAE, version 5.0, grade 3 - 4
Measurement of geriatric recommendations | at 3, 6 and 12 months since the start of systemic therapy
  Number of geriatric recommendations and adherence of geriatric recommendations (= geriatric interventions)
Measurement of actions undertaken | at 3, 6 and 12 months since the start of systemic therapy
  Number of actions undertaken within the geriatric interventions and adherence to actions undertaken (= patient compliance) defined as the degree to which a patient correctly follows the actions undertaken within the geriatric interventions.
Overall Survival | over 2 year follow-up since the start of systemic therapy
  the length of time from the start of treatment and death from any cause
Number of patients with premature interruption of systemic therapy | over 1 year follow up since the start of the systemic therapy
  Premature interruption of systemic therapy is defined as the complete discontinuation of the systemic therapy the patient receives in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, prof. dr., Principal Investigator — adjunct head of clinic
Locations (1):
- UZ Gasthuisberg Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenis C, Peeters L, Laethem L, De Cock J, Compte N, Flamaing J, Milisen K, Fagard K, Lobelle JP, Laenen A, Decoster L, Wildiers H. Effectiveness of comprehensive geriatric assessment with extensive patient coaching for improving quality of life in older patients with solid tumours receiving systemic therapy (G-oncoCOACH): a multicentre randomised controlled trial. Lancet Healthy Longev. 2025 Aug;6(8):100743. doi: 10.1016/j.lanhl.2025.100743. Epub 2025 Aug 13. PMID 40818480